CLINICAL TRIAL: NCT04898335
Title: TENDyne European expeRience Registry
Acronym: TENDER
Status: Recruiting | Type: Observational
Sponsor: LMU Klinikum (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Jörg Hausleiter, Prof. Dr. med. Jörg Hausleiter, LMU Klinikum
Other Study IDs: 21-0110
Record Dates: First submitted 2021-04-30; First posted 2021-05-24 (Actual); Last update posted 2021-05-24 (Actual); Status verified 2021-05

CONDITIONS: Mitral Regurgitation
Keywords: mitral regurgitation; Tendyne; transcatheter mitral valve replacement
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Tendyne: all patients treated with a Tendyne Mitral Valve System
  Interventions: Device: Tendyne Mitral Valve System

INTERVENTIONS:
Device: Tendyne Mitral Valve System — Tendyne Mitral Valve System for mitral valve disease in a commercial setting

SUMMARY:
TENDER is a multicenter, single-device, retrospective and prospective, observational study to assess safety and efficacy of the Tendyne Mitral Valve System in a real-world population.

DETAILED DESCRIPTION:
Mitral regurgitation (MR) is a common disease and is associated with high morbidity and mortality if left untreated. Due to age and comorbidities, patients are often ineligible for surgical repair or replacement. Over the last years, transcatheter systems have been introduced as an alternative therapeutic approach. The Tendyne Mitral Valve System (Abbott Vascular, Roseville, Minnesota) is a transcatheter transapical, self-expanding valve prosthesis for mitral valve replacement. A recent study has proven safety and feasibilty of the system, leading to commercial approvement (CE mark). However, data on real world experience with the system are not available.

TENDER is a multicenter, single-device, retrospective and prospective, observational study. Objectives of the study are 1) to assess early outcomes, including safety and efficacy, in patients treated with the Tendyne Mitral Valve System for severe MR at 30 days, 2) to assess clinical outcomes in patients treated with the Tendyne Mitral Valve System for severe MR at 1 year and 3 year follow-up, and 3) to identify echocardiographic and CT-based anatomic predictors associated with outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated with the Tendyne Mitral Valve System for mitral valve disease in a commercial setting
* Patients providing written informed consent in compliance with the protocol, the ICH-GCP and all national legal and regulatory requirements

Exclusion Criteria:

* Patients not providing written informed consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All consecutive patients undergoing Implantation of Tendyne Mitral Valve System at the participating centres.
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of procedural success | 30 days
  Device success (structural and functional); absence of death, stroke, life-threatening bleeding, major vascular or cardiac structural complications, acute kidney injury, myocardial infarction, heart failure and valve-related dysfunction requiring repeat procedure

SECONDARY OUTCOMES:
Rate of peri-procedural myocardial infarction | 1 day
  Myocardial infarction during the index procedure
Rate of conversion to open-heart surgery | 1 day
  Conversion to open-heart surgery during the index procedure
Rate of cardiac tamponade | 1 day
  Cardiac Tamponade during the index procedure
Rate of procedural mortality | 1 day
  Death during the index procedure
Rate of technical success (cumulative endpoint according to MVARC) | 1 day
  Absence of procedural mortality, successful access, delivery and retrieval of the delivery system, successful deployment and positioning, freedom from emergency surgery) Device success (according to MVARC): absence of procedural mortality or stroke, proper placement and positioning, freedom from unplaned procedure related to the device or access, continued safety and performance of the device (no structural or functional failure, no technical complications, reduction of MR ≤ 2+ and mitral valve gradient < 5 mmHg)
Rate of device success (cumulative endpoint according to MVARC) | 30 days, 1 year and 3 years
  Absence of procedural mortality or stroke, proper placement and positioning, freedom from unplaned procedure related to the device or access, continued safety and performance of the device (no structural or functional failure, no technical complications, reduction of MR ≤ 2+ and mitral valve gradient < 5 mmHg)
New York Heart Association (NYHA) functional class | 30 days, 1 year and 3 years
  class I - IV
6-minute walk distance (6MWD) | 30 days, 1 year and 3 years
  in m
BNP/NT-proBNP level | 30 days, 1 year and 3 years
  in pg/ml
Mitral regurgitation severity grade | 30 days, 1 year and 3 years
  grade 0/1+/2+/3+/4+
Left and right ventricular dimensions | 30 days, 1 year and 3 years
  left/right ventricular end-diastolic/-systolic diameter (in mm)
Left ventricular function | 30 days, 1 year and 3 years
  LVEF in percent
Right ventricular function | 30 days, 1 year and 3 years
  TAPSE in mm
Pulmonary artery pressure | 30 days, 1 year and 3 years
  in mmHg
Tricuspid regurgitation severity grade | 30 days, 1 year and 3 years
  grade 1-5
Transprosthetic gradient | 30 days, 1 year and 3 years
  in mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Hausleiter, MD, Principal Investigator — LMU Klinikum Munich
Locations (30):
- Austria (2):
  - Universitaetsklinikum Linz, Linz
  - Universitaetsklinikum Wien, Vienna
- UZ Leuven, Leuven, Belgium
- France (4):
  - CHU de Bordeaux, Bordeaux
  - CHU de Lille, Lille
  - CHU Rennes, Rennes
  - Clinique Pasteur, Toulouse
- Germany (12):
  - Herz- und Diabeteszentrum NRW, Bad Oeynhausen
  - Deutsches Herzzentrum Berlin, Berlin
  - Universitaetsklinikum Bonn, Bonn
  - Universitaetsklinikum Koeln, Cologne
  - Universitätsklinikum Frankfurt, Frankfurt
  - UKE Hamburg, Hamburg
  - Herzentrum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - DHZ München, Münich
  - Universitaetsklinikum Regensburg, Regensburg
  - Robert-Bosch-Krankenhaus Stuttgart, Stuttgart
  - Universitaetsklinikum Tuebingen, Tübingen
- Italy (2):
  - ICH - Istituto Clinico Humanitas, Milan
  - University Hospital of Pisa, Pisa
- University hospital Oslo, Oslo, Norway
- Spain (4):
  - Puerto de Hierro Madrid, Madrid
  - University hospital Madrid, Madrid
  - Hospital Clinico Valladolid, Valladolid
  - University Hospital of Vigo, Vigo
- Karolinska University Stockholm, Stockholm, Sweden
- Switzerland (2):
  - Universitaetsspital Basel, Basel
  - Inselspital Bern, Bern
- Royal Brompton London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hell MM, Wild MG, Baldus S, Rudolph T, Treede H, Petronio AS, Modine T, Andreas M, Coisne A, Duncan A, Franco LN, Praz F, Ruge H, Conradi L, Zierer A, Anselmi A, Dumonteil N, Nickenig G, Pinon M, Barth S, Adamo M, Dubois C, Torracca L, Maisano F, Lurz P, von Bardeleben RS, Hausleiter J; TENDER Investigators. Transapical Mitral Valve Replacement: 1-Year Results of the Real-World Tendyne European Experience Registry. JACC Cardiovasc Interv. 2024 Mar 11;17(5):648-661. doi: 10.1016/j.jcin.2023.12.027. Epub 2024 Feb 21. PMID 38385922